CLINICAL TRIAL: NCT01803789
Title: Single Versus Double Kirschner Wires for Intramedullary Fixation of Metacarpal V Fractures
Acronym: 1-2-KiWI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medicine Greifswald (Other)
Collaborators: Deutsche Arthrose-Hilfe (Other)
Responsible Party: Principal Investigator, Prof. Dr. Andreas Eisenschenk, Prof. Dr., University Medicine Greifswald
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1-2-KiWI
Record Dates: First submitted 2013-03-01; First posted 2013-03-04 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-11

CONDITIONS: Fracture of Metacarpal Bone
Keywords: Metacarpal V Fractures; Single Kirschner Wires; Double Kirschner Wires
MeSH Terms: interventions — Bone Wires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Single Kirschner Wire (Active Comparator): Antegrade intramedullary fixation of with a single Kirschner wire.
  Interventions: Device: Single Kirschner Wire
- Double Kirschner Wire (Active Comparator): Antegrade intramedullary fixation with double Kirschner wire.
  Interventions: Device: Double Kirschner Wire

INTERVENTIONS:
Device: Single Kirschner Wire
  Arms: Single Kirschner Wire
Device: Double Kirschner Wire
  Arms: Double Kirschner Wire

SUMMARY:
Metacarpal V fractures are injuries of the upper extremities. They occur frequently, primarily in young adults.These fractures are caused by falling on the fist, sports accidents and direct or indirect forces.

Surgical intervention is necessary for fractures with a strong palmar angulation of the metacarpal bone or rotational deformity of the small finger. Due to the absence of guideline recommendations decisions about therapy are made taking into account logistical aspects, available hardware, individual expertise and preferences. The objective of the study is to compare the advantages and disadvantages of single versus double Kirschner wires for intramedullary fixation of metacarpal V fractures in order to standardize national therapy procedures.

Primary hypothesis:

In the surgical therapy of the dislocated and/or rotational deformed metacarpal V neck fracture, osteosynthesis with a single Kirschner wire is not inferior to osteosynthesis with a double Kirschner wire with regard to the functional outcome after 6 month, as measured with the Disabilities of the Arm, Shoulder and Hands Score (DASH).

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥18 years with a metacarpal V neck fracture with a palmar angulation and/or shortening and /or rotational deformity as determined on radiological diagnosis
* Trauma within 10 days before appearing in the study centre
* No specific medical treatment before
* Ability to fully understand the character and implications of the clinical trial
* Written or oral (in case of an injury of the dominant hand, if so attested by witnesses)consent

Exclusion Criteria:

* Indications for conservative therapy
* Patient is not suitable for anaesthesia
* Other physical conditions or characteristics which made surgical interventions inappropriate or to risky (e.g. open fractures, polytrauma, pregnancy, acute infections, pathological fractures)
* Prior participation in this study (e.g. injury of the contralateral hand) or participation in other interventional studies with the same objective
* Physical or mental diseases which makes the consequent participation in diagnostic, therapy and the follow-up-examinations unlikely
* Lacking language skills

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 292 (Actual)
Dates: Start 2013-05; Primary Completion 2017-06 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Differences in functional outcome of the therapy with single or double Kirschner wires measured with the DASH score | 6 months after randomisation

SECONDARY OUTCOMES:
Malposition or angulation in the frontal and sagittal planes of max. 5° | 6 months after randomisation
Shortening of the metacarpus >2mm | 6 months after randomisation
Palmar angulation >30° | 6 months after randomisation
Non-union/Pseudarthrosis | 6 months after randomisation
Limitation of fist closure | 6 months after randomisation
Flexion or extension lag | 6 months after randomisation
Pain intensity <10 points (VAS) | 6 months after randomisation
Duration of surgical intervention | 6 months after randomisation
Rate of re-interventions | 6 months after randomisation
Rate of infections | 6 months after randomisation
Rate of perforation/dislocation/break of the fracture fixation devices | 6 months after randomisation
Duration of inability to work | 6 months after randomisation

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Eisenschenk, Prof. Dr., Principal Investigator — University Medicine Greifswald
Locations (12):
- Germany (12):
  - University Medicine Greifswald, Greifswald, Mecklenburg-Vorpommern
  - Sana Clinical Centre Lichtenberg, Berlin
  - Vivantes Hospital Am Urban, Berlin
  - Trauma Hospital Berlin, Berlin
  - University Medicine Düsseldorf, Düsseldorf
  - District Hospital Gummersbach, Gummersbach
  - BG Kliniken Bergmannstrost, Halle
  - Berufsgenossenschaftliches Unfallkrankenhaus Hamburg, Hamburg
  - University Medicine Hamburg-Eppendorf, Hamburg
  - Berufsgenossenschaftliches Unfallkrankenhaus Ludwigshafen, Ludwigshafen
  - University Medicine Rostock, Rostock
  - Municipal Clinic Solingen, Solingen

IPD SHARING:
Plan to Share IPD: No